CLINICAL TRIAL: NCT01609543
Title: Open Label Study of Erlotinib (Tarceva®) as Single Agent First Line Treatment of Patients With Locally Advanced or Metastatic Lung Adenocarcinoma With Activating Epidermal Growth Factor Receptor (EGFR) Mutations
Brief Title: A Study of Tarceva (Erlotinib) in First Line in Patients With Locally Advanced or Metastatic Lung Adenocarcinoma With EGFR Mutations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML27880; 2011-002168-26 (EudraCT Number)
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg orally daily, until disease progression, unacceptable toxicity or withdrawal due to any reason

SUMMARY:
This open-label, non-randomized, one-arm study will evaluate the safety and efficacy of Tarceva (erlotinib) as single-agent first-line treatment in patients with locally advanced or metastatic non-small cell lung cancer who show epidermal growth factor receptor (EGFR) activating mutations. Patients will receive Tarceva 150 mg orally daily until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically documented, inoperable, locally advanced, recurrent or metastatic (Stage IIIB or Stage IV) lung adenocarcinoma
* Non-small cell lung cancer with an EGFR activating mutation
* Patients must have evidence of disease, but measurable disease is not mandatory
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate renal and liver function

Exclusion Criteria:

* Prior chemotherapy or other systemic anti-cancer treatment. Neoadjuvant/adjuvant chemotherapy is allowed if completed within 6 months prior to enrolment. Prior radiochemotherapy is allowed if completed more than 6 months before start of study treatment
* Prior therapy with systemic anti-tumour therapy with HER1/EGFR inhibitors
* Any other malignancies within 5 years, except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin carcinoma
* Brain metastasis or spinal cord compression not yet definitely treated with surgery and/or radiation
* Patients unable to take oral medication or requiring intravenous alimentation, with prior surgical procedures affecting absorption or active peptic ulcer disease
* Any significant ophthalmologic abnormality, especially those likely to increase the risk of corneal epithelial lesions; the use of contact lenses is not recommended during the study
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Hungary (14):
  - Budapest
  - Debrecen
  - Deszk
  - Farkasgyepű
  - Gyula
  - Mátraháza
  - Mosonmagyaróvar
  - Nyíregyháza
  - Pécs
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Törökbálint
- Riga, Latvia
- Turkey (Türkiye) (4):
  - Ankara
  - Antalya
  - Edirne
  - Istanbul

REFERENCES:
- [Derived] Markoczy Z, Sarosi V, Kudaba I, Galffy G, Turay UY, Demirkazik A, Purkalne G, Somfay A, Papai-Szekely Z, Raso E, Ostoros G. Erlotinib as single agent first line treatment in locally advanced or metastatic activating EGFR mutation-positive lung adenocarcinoma (CEETAC): an open-label, non-randomized, multicenter, phase IV clinical trial. BMC Cancer. 2018 May 25;18(1):598. doi: 10.1186/s12885-018-4283-z. PMID 29801465

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 651 participants were screened and among them 62 participants were enrolled in the study.
Groups:
- Erlotinib Hydrochloride: Participants received a single 150 milligrams (mg) oral dose of erlotinib hydrochloride (Tarceva) tablet daily from Day 1 until disease progression, death, unacceptable toxicity or consent withdrawal, whichever occurred first up to 34 months.
Period: Overall Study
Arm/Group | Erlotinib Hydrochloride
Started | 62
Completed | 20
Not Completed | 42
Not completed — Disease Progression | 28
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants.
Groups:
- Erlotinib Hydrochloride: Participants received a single 150 mg oral dose of erlotinib hydrochloride tablet daily from Day 1 until disease progression, death, unacceptable toxicity or consent withdrawal, whichever occurred first up to 34 months.
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.69 (10.562)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as median time from the first dose of study treatment to the first documentation of objective tumor progression (according to Response Evaluation Criteria in Solid Tumours [RECIST] version 1.1) or to death due to any cause, whichever occurred first. Progressive Disease (PD) was defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression. Median and the 95% confidence interval were estimated using Kaplan-Meier survival methodology.
Time Frame: Baseline to progressive disease or death (up to 34 months)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Erlotinib Hydrochloride: Participants received a single 150 mg oral dose erlotinib hydrochloride tablet daily from Day 1 until disease progression, death, unacceptable toxicity, or consent withdrawal, whichever occurred first up to 34 months.
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 62
Months | 12.846 [9.901 to 15.791]

2. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR)
Description: BOR was defined as best tumor response (as per RECIST version 1.1) recorded for a participant during the study. Complete Response (CR): disappearance of all target and non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (less than [<] 10 millimeters [mm] short axis). Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Baseline to progressive disease or death (up to 34 months)
Population: ITT population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 62
Percentage of Participants
  CR | 1.8
  PR | 64.3
  SD | 32.1
  PD | 1.8

3. Secondary Outcome: Percentage of Participants Who Were Alive at 1 Year
Time Frame: 1 Year (12 months)
Population: ITT population. Here, number of participants analyzed signifies those participants who were evaluable for this outcome.
Measure: Number; unit: Percentage of Participants
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 40
Percentage of Participants | 82.5

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last dose of study medication (up to 34 months)
Arm/Group | Erlotinib Hydrochloride
Serious Adverse Events (participants affected / at risk) | 26/62
Other Adverse Events (participants affected / at risk) | 49/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Hydrochloride (N=62)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Ileus Paralytic (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden Cardiac Death (General disorders) | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Liver Injury (Hepatobiliary disorders) | 2
Pneumonia (Infections and infestations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Liver Function Test Abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance Disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Renal Failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Rash Generalised (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Hydrochloride (N=62)
Anaemia (Blood and lymphatic system disorders) | 5
Growth of Eyelashes (Eye disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 5
Conjunctivitis (Infections and infestations) | 6
Blood Alkaline Phosphatase Increased (Investigations) | 5
Weight Decreased (Investigations) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.